CLINICAL TRIAL: NCT03874598
Title: Effectiveness of Ear Acupuncture to Improve Insomnia in Women With Breast Cancer: a Randomized Controlled Trial
Brief Title: Effectiveness of Ear Acupuncture to Improve Insomnia in Women With Breast Cancer
Acronym: EOMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: Karl and Veronica Carstens Foundation (Other)
Responsible Party: Principal Investigator, Dr. med. Petra Voiss, MD, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-8214-BO; KVC 0/100/2018 (Other Grant/Funding Number: Karl und Veronica Carstens-Foundation)
Record Dates: First submitted 2019-03-13; First posted 2019-03-14 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Breast Neoplasm
Keywords: Sleep Initiation and Maintenance Disorders; Acupuncture, Ear; Cytokines; Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms; Sleep Initiation and Maintenance Disorders | interventions — Acupuncture, Ear

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ear acupuncture (Experimental)
  Interventions: Procedure: Ear acupuncture
- Psychoeducation (Active Comparator)
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Procedure: Ear acupuncture — Patients in the intervention group are treated twice a week for five weeks using semi-standardized ear acupuncture.
  Arms: Ear acupuncture
Behavioral: Psychoeducation — Patients of the control group receive a 1,5 h psychoeducation group concerning sleep improving behaviour.
  Arms: Psychoeducation

SUMMARY:
The aim of this clinical study is to investigate the extent to which ear acupuncture has an effect on insomnia in women with breast cancer. It will be investigated whether changes in sleep quality, fatigue, quality of life, stress, and psychological well-being can be achieved. In addition, a proinflammatory cytokine will be meassured.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosed non-metastatic breast CAs (TNM stage I-III)
* Existing insomnia (difficulty falling asleep or sleeping through on at least 3 days per week for at least 3 months) according to the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders (DSM 5).
* willingness to participate in the study (at least 8 out of 10 treatments)
* Signed informed consent

Exclusion Criteria:

* Ongoing or planned chemotherapy, radiation, follow-up treatment or reconstructive plastic surgery during the study period
* Severe physical or psychopharmacologically treated psychiatric comorbidity that prevents a patient from participating in the study
* Pregnancy
* Participation in other clinical trials with behavioural, psychological or complementary medical interventions during the study period
* Regular use of barbiturates, antidepressants or other sleep-inducing drugs, drug abusus, alcoholism

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Sleep Quality | week 0
  Pittsburgh Sleep Quality Index (PSQI). The PSQI contains 19 self-assessment questions and 5 questions rated by the bed-partner or roommate. The 5 questions rated by the bed-partner or roommate are only used as clinical information and not included in qualitative analysis. The question whether a bed-partner or roommate is present is not included in qualitative analysis as well. The 18 self-assessment items are used to evaluate the sleep quality on 7 domains over the last month (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, and sleep disturbances, use of sleep medication, and daytime dysfunction). Scoring of the answers is based on a scale from 0 to 3, whereby 3 reflects the negative extreme on a Likert Scale. The total score is generated by the summation of the component scores and can vary from 0 to 21, with a higher score corresponding to a reduced sleep quality. A cut-off score of 5 indicates a "poor" sleeper.
Sleep Quality | week 5
  Pittsburgh Sleep Quality Index (PSQI). The PSQI contains 19 self-assessment questions and 5 questions rated by the bed-partner or roommate. The 5 questions rated by the bed-partner or roommate are only used as clinical information and not included in qualitative analysis. The question whether a bed-partner or roommate is present is not included in qualitative analysis as well. The 18 self-assessment items are used to evaluate the sleep quality on 7 domains over the last month (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, and sleep disturbances, use of sleep medication, and daytime dysfunction). Scoring of the answers is based on a scale from 0 to 3, whereby 3 reflects the negative extreme on a Likert Scale. The total score is generated by the summation of the component scores and can vary from 0 to 21, with a higher score corresponding to a reduced sleep quality. A cut-off score of 5 indicates a "poor" sleeper.

SECONDARY OUTCOMES:
Quality of Life in cancer patients | week 0
  Functional Assessment Of Cancer Therapy - Breast Cancer (FACT-B)
Quality of Life in cancer patients | week 5
  Functional Assessment Of Cancer Therapy - Breast Cancer (FACT-B)
Quality of Life in cancer patients | week 17
  Functional Assessment Of Cancer Therapy - Breast Cancer (FACT-B)
Quality of Life in cancer patients | week 29
  Functional Assessment Of Cancer Therapy - Breast Cancer (FACT-B)
Fatigue | week 0
  Functional Assessment Of Chronic Illness Therapy - Fatigue (FACIT-F)
Fatigue | week 5
  Functional Assessment Of Chronic Illness Therapy - Fatigue (FACIT-F)
Fatigue | week 17
  Functional Assessment Of Chronic Illness Therapy - Fatigue (FACIT-F)
Fatigue | week 29
  Functional Assessment Of Chronic Illness Therapy - Fatigue (FACIT-F)
Psychological well-being | week 0
  Hospital Anxiety and Depression Scale (HADS). It measures the 2 dimensions anxiety and depression. Scores range from 0 to 21 with higher values indicate higher distress. Values of >8 indicate potential subclinical anxiety or depressive disorders.
Psychological well-being | week 5
  Hospital Anxiety and Depression Scale (HADS). It measures the 2 dimensions anxiety and depression. Scores range from 0 to 21 with higher values indicate higher distress. Values of >8 indicate potential subclinical anxiety or depressive disorders.
Psychological well-being | week 17
  Hospital Anxiety and Depression Scale (HADS). It measures the 2 dimensions anxiety and depression. Scores range from 0 to 21 with higher values indicate higher distress. Values of >8 indicate potential subclinical anxiety or depressive disorders.
Psychological well-being | week 29
  Hospital Anxiety and Depression Scale (HADS). It measures the 2 dimensions anxiety and depression. Scores range from 0 to 21 with higher values indicate higher distress. Values of >8 indicate potential subclinical anxiety or depressive disorders.
Stress | week 0
  Perceived Stress Scale (PSS). Perceived stress will be assessed by the 10-item version of the PSS, rated for the past month on a 5-point rating scale. For the summed items (range from 0 to 40) a higher total score indicates greater stress.
Stress | week 5
  Perceived Stress Scale (PSS). Perceived stress will be assessed by the 10-item version of the PSS, rated for the past month on a 5-point rating scale. For the summed items (range from 0 to 40) a higher total score indicates greater stress.
Stress | week 17
  Perceived Stress Scale (PSS). Perceived stress will be assessed by the 10-item version of the PSS, rated for the past month on a 5-point rating scale. For the summed items (range from 0 to 40) a higher total score indicates greater stress.
Stress | week 29
  Perceived Stress Scale (PSS). Perceived stress will be assessed by the 10-item version of the PSS, rated for the past month on a 5-point rating scale. For the summed items (range from 0 to 40) a higher total score indicates greater stress.
Adverse Events | week 5
  Number of patients with adverse events and type of the adverse event
Adverse Events | week 17
  Number of patients with adverse events and type of the adverse event
Change in proinflammatory cytokine | week 0
  Interleukin-6
Change in proinflammatory cytokine | week 5
  Interleukin-6
Expectation | week 0
  Visual Analogue Scale (VAS). The Visual Analogue Scale is a continuous measurement device on which the degree of agreement is indicated by a cross between two end points. We define the end points of the Visual Analalogue Scale for expectations concerning treatment as "expecting the treatment to be not sucessfull at al" and "expecting the treatment to be extremely successful.
Sleep Quality | week 17
  Pittsburgh Sleep Quality Index (PSQI). The PSQI contains 19 self-assessment questions and 5 questions rated by the bed-partner or roommate. The 5 questions rated by the bed-partner or roommate are only used as clinical information and not included in qualitative analysis. The question whether a bed-partner or roommate is present is not included in qualitative analysis as well. The 18 self-assessment items are used to evaluate the sleep quality on 7 domains over the last month (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, and sleep disturbances, use of sleep medication, and daytime dysfunction). Scoring of the answers is based on a scale from 0 to 3, whereby 3 reflects the negative extreme on a Likert Scale. The total score is generated by the summation of the component scores and can vary from 0 to 21, with a higher score corresponding to a reduced sleep quality. A cut-off score of 5 indicates a "poor" sleeper.
Sleep Quality | week 29
  Pittsburgh Sleep Quality Index (PSQI). The PSQI contains 19 self-assessment questions and 5 questions rated by the bed-partner or roommate. The 5 questions rated by the bed-partner or roommate are only used as clinical information and not included in qualitative analysis. The question whether a bed-partner or roommate is present is not included in qualitative analysis as well. The 18 self-assessment items are used to evaluate the sleep quality on 7 domains over the last month (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, and sleep disturbances, use of sleep medication, and daytime dysfunction). Scoring of the answers is based on a scale from 0 to 3, whereby 3 reflects the negative extreme on a Likert Scale. The total score is generated by the summation of the component scores and can vary from 0 to 21, with a higher score corresponding to a reduced sleep quality. A cut-off score of 5 indicates a "poor" sleeper.

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Dobos, Prof. MD, Study Director — University of Duisburg Essen
Locations (1):
- Kliniken Essen-Mitte, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No